CLINICAL TRIAL: NCT01097954
Title: A Prospective Study Measuring Exhaled Nitric Oxide in Exercise-Induced Asthma
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 146548
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Exercise Induced Asthma
Keywords: Exercise induced asthma; Exercise induced bronchospasm; exhaled Nitric Oxide
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Exercise induced bronchospasm (EIB), also known as exercise induced asthma (EIA) is a transient obstruction to airflow triggered by exertion.

It is now a well known identity, center of discussion in recent years, particularly in the athletes' world. It is more common in asthmatic individuals (regardless of severity of disease), but it is also seen in otherwise healthy subjects, leading to the general consensus that the pathophysiology is different than asthma.

The concentration of exhaled nitric oxide (FeNO) in various airway & respiratory disorders, particularly asthma, has been deeply studied. Its use for noninvasive monitoring of asthma control (reflecting airway eosinophilic inflammation) is being closely examined and put into clinical practice. FeNO is significantly elevated in asthma. Elevated FeNO levels have also been noted in patients hospitalized with a COPD exacerbation, acidosis, rhinitis, bronchiectasis, active pulmonary sarcoidosis, active fibrosing alveolitis, and acute lung allograft rejection. Decreased FeNO levels have been seen in patients with primary ciliary dyskinesia, cystic fibrosis, PiZZ phenotype-related alpha-1 antitrypsin deficiency, and pulmonary hypertension

Two studies have addressed the variations on FeNO after EIB and they had contradictory results. Scollo et al. found no change in FeNO in either healthy or asthmatic children after a 6-min of vigorous exertion in an exercise laboratory when they studied 24 asthmatic and 18 control children. Terada et al. reported, for 39 subjects, a decrease in FeNO in subjects with EIB and an increase in healthy controls.

It is well accepted that the pathophysiology of exercise induced bronchospasm it is not similar to that of asthma. Certainly the inflammation in the airway does not appear to be eosinophilic. Understanding the disease mechanism is a key factor to adequately manage it.

This will be a prospective study measuring online exhaled nitric oxide involving children 8 to 21 years old. The study group will include any children coming for a pulmonary exercise test in the exercise laboratory located in the Pediatric Pulmonary Division office.

The study will be conducted from the fall of 2009 until the spring of 2011. The change in the FeNO measurement will be correlated with the change in % predicted FEV1. We will consider significant a decrease in FEV1 post exercise of 15% and/or decrease on FEF25-75 of 20% that will persist until 15 minutes after completing exercise.

We will also record any symptoms reported by the subject during or after the test.

An exercise test is a standard of care when suspecting exercise-induced asthma. The subjects and their parents coming for exercise test will be offered the opportunity to participate in the study.

The subject will come for the exercise test and will perform spirometry and FeNO measurement prior to start the test. According to our exercise laboratory protocol 1 minute of warm up at a low speed, followed by 6 minutes of high speed (enough to increase heart rate to 90% predicted or more) and 3 minutes of cool down at a low speed will be performed.

Then spirometry will be repeated at 3, 5, 10 and 15 minutes and FeNO measurement will be taken at 5, 10 and 15 minutes.

We will analyze the data to find if there is any significant change in FeNO measurements after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 8-21 years of age coming for an exercise stress test at the Pediatric Pulmonary office at Winthrop University Hospital with symptoms consistent with exercise induced asthma

Exclusion Criteria:

* Do not meet the diagnosis of exercise induced asthma
* Can not perform a sub-maximal exercise test on a treadmill due to orthopedic limitations
* Are under age 8 years old and will not be able to perform an exercise test and/or nitric oxide test
* Have severe persistent asthma with baseline increased levels of nitric oxide
* Diagnosed with any chronic lung disease, hypertension, heart failure, pulmonary hypertension, primary ciliary dyskinesia, bronchiectasis, alveolitis, lung transplant rejection, pulmonary sarcoidosis, chronic cough (i.e. greater four weeks), systemic sclerosis, hypersensitivity, cystic fibrosis, HIV, sickle cell anemia, cardiac pulmonary bypass, liver cirrhosis, alpha-1 anti-trypsin disease and interstitial lung

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subject with symptoms consistent with exercise induced asthma
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Variations in the fraction of exhaled nitric oxide in subjects with exercise induced asthma | 1 year
  The exhaled Nitric Oxide (FeNO) will be measured before the exercise test and at 5, 10 and 15 min after completion of the exercise to detect variations in the value

SECONDARY OUTCOMES:
Correlation between level of FeNO and reduction in FEV1 | 1 year
  Variations in the FeNO will be compared to FEV1 changes to see if they correlate
Correlation between level of FeNO and severity of symptoms | 1 year
  Variations in FeNO will be correlated with symptoms reported

CONTACTS AND LOCATIONS:
Overall Officials: Melodi Pirzada, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Anderson SD, Kippelen P. Airway injury as a mechanism for exercise-induced bronchoconstriction in elite athletes. J Allergy Clin Immunol. 2008 Aug;122(2):225-35; quiz 236-7. doi: 10.1016/j.jaci.2008.05.001. Epub 2008 Jun 12. PMID 18554705
- [Background] Sue-Chu M, Larsson L, Bjermer L. Prevalence of asthma in young cross-country skiers in central Scandinavia: differences between Norway and Sweden. Respir Med. 1996 Feb;90(2):99-105. doi: 10.1016/s0954-6111(96)90206-1. PMID 8730329
- [Background] Baraldi E, de Jongste JC; European Respiratory Society/American Thoracic Society (ERS/ATS) Task Force. Measurement of exhaled nitric oxide in children, 2001. Eur Respir J. 2002 Jul;20(1):223-37. doi: 10.1183/09031936.02.00293102. PMID 12166573
- [Background] Ricciardolo FL, Sterk PJ, Gaston B, Folkerts G. Nitric oxide in health and disease of the respiratory system. Physiol Rev. 2004 Jul;84(3):731-65. doi: 10.1152/physrev.00034.2003. PMID 15269335
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] Bult H, Boeckxstaens GE, Pelckmans PA, Jordaens FH, Van Maercke YM, Herman AG. Nitric oxide as an inhibitory non-adrenergic non-cholinergic neurotransmitter. Nature. 1990 May 24;345(6273):346-7. doi: 10.1038/345346a0. PMID 1971425
- [Background] Anderson SD, Daviskas E. The airway microvasculature and exercise induced asthma. Thorax. 1992 Sep;47(9):748-52. doi: 10.1136/thx.47.9.748. PMID 1440473
- [Result] Scollo M, Zanconato S, Ongaro R, Zaramella C, Zacchello F, Baraldi E. Exhaled nitric oxide and exercise-induced bronchoconstriction in asthmatic children. Am J Respir Crit Care Med. 2000 Mar;161(3 Pt 1):1047-50. doi: 10.1164/ajrccm.161.3.9905043. PMID 10712361
- [Result] Buchvald F, Hermansen MN, Nielsen KG, Bisgaard H. Exhaled nitric oxide predicts exercise-induced bronchoconstriction in asthmatic school children. Chest. 2005 Oct;128(4):1964-7. doi: 10.1378/chest.128.4.1964. PMID 16236842
- [Result] Terada A, Fujisawa T, Togashi K, Miyazaki T, Katsumata H, Atsuta J, Iguchi K, Kamiya H, Togari H. Exhaled nitric oxide decreases during exercise-induced bronchoconstriction in children with asthma. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1879-84. doi: 10.1164/ajrccm.164.10.2009105. PMID 11734440
- [Result] Nishio K, Odajima H, Motomura C, Nakao F, Nishima S. Exhaled nitric oxide and exercise-induced bronchospasm assessed by FEV1, FEF25-75% in childhood asthma. J Asthma. 2007 Jul-Aug;44(6):475-8. doi: 10.1080/02770900701424090. PMID 17654135
- [Result] Garcia-Rio F, Ramirez M, Mediano O, Lores V, Rojo B, Villasante C, Villamor J. Exhaled nitric oxide and airway caliber during exercise-induced bronchoconstriction. Int J Sports Med. 2006 Nov;27(11):905-10. doi: 10.1055/s-2006-923775. PMID 17120347